CLINICAL TRIAL: NCT01048736
Title: Investigating Fitness Interventions in the Elderly (INFINITE)
Acronym: INFINITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00008292; 40010566 (Other Grant/Funding Number: National Heart Lung and Blood Institute)
Record Dates: First submitted 2010-01-11; First posted 2010-01-14 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2018-07

CONDITIONS: Obesity; Older Adults; Sedentary
Keywords: obesity; exercise; intensity; weight loss; diet
MeSH Terms: conditions — Obesity; Sedentary Behavior; Motor Activity; Weight Loss | interventions — Exercise; Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise (Active Comparator): All treatment groups will receive 4d/wk of exercise
  Interventions: Behavioral: Exercise Only
- Exercise + Diet (-250 kcal/d deficit) (Experimental): Exercise 4d/wk with moderate caloric restriction (-250 kcal/d deficit) designed for low fat loss (EX+Low CR; ~4.5 kg weight loss),
  Interventions: Behavioral: Exercise + Diet
- Exercise + Diet (-600 kcal/d deficit) (Experimental): Exercise 4d/wk with intensive caloric restriction (-600 kcal/d deficit) designed for high fat loss (EX+High CR; ~10.9 kg weight loss)
  Interventions: Behavioral: Exercise + Diet

INTERVENTIONS:
Behavioral: Exercise Only — 4 d/wk of aerobic exercise
  Other Names: EX
  Arms: Exercise
Behavioral: Exercise + Diet — Exercise 4d/wk with moderate caloric restriction (-250 kcal/d deficit) designed for low fat loss (EX+Low CR; ~4.5 kg weight loss).
  Other Names: EX+Low CR
  Arms: Exercise + Diet (-250 kcal/d deficit)
Behavioral: Exercise + Diet — Exercise 4d/wk with intensive caloric restriction (-600 kcal/d deficit) designed for high fat loss (EX+High CR; ~10.9 kg weight loss)
  Other Names: EX+ High CR
  Arms: Exercise + Diet (-600 kcal/d deficit)

SUMMARY:
Aging is associated with declines in aerobic capacity, exercise tolerance, and functional endurance that lead to physical disability and loss of independence. Furthermore, the existing high prevalence of obesity in the elderly is greatly exacerbating these aging-related declines in function. To date, regular exercise is the only known therapy to consistently improve aerobic function, and perhaps delay the onset of disability. Although aerobic exercise training does benefit both aerobic capacity and endurance even in obese persons, some data show that the maximal efficacy of exercise for improving aerobic function is blunted by obesity. In addition, our preliminary data show a potential dose-response benefit of concomitant fat loss on exercise-induced improvements in aerobic function. Thus, combining an exercise intervention with caloric restriction resulting in fat loss may be more efficacious for improving aerobic function than exercise alone in obese elderly, a population at high risk for disability. The purpose of this study is to determine whether the amount of fat loss (achieved through controlled underfeeding) affects the magnitude of improvement in aerobic function (maximal aerobic capacity and endurance) in response to a standardized exercise training stimulus that follows current recommendations for older persons.

DETAILED DESCRIPTION:
Design Overview:

Phase 1 involves recruitment and screening followed by baseline research testing (Phase 2). Next, subjects will be randomly assigned to one of three 5-month treatments (Phase 3): exercise and high-caloric restriction diet, exercise and low-caloric restriction diet, or exercise only. Subjects will complete follow-up testing after their 5 month intervention.

Interventions:

Dietary interventions: All participants will be randomly assigned to an exercise intervention with either no dietary intervention (EX Only), or 1 of 2 hypocaloric controlled diets: 1) -250 kcal/day deficit for low fat loss (EX+LOW CR) or 2) -600 kcal/day deficit for high fat loss (EX+HIGH CR) for 20 weeks.

All meals are prepared individually after participants choose from a hypocaloric menu designed by the RD to provide a balanced, healthy diet. The calorie level assigned for each person will provide him/her with an absolute daily caloric deficit consistent with their group assignment (-600 or -250 kcals/day). Individual calorie levels will be prescribed to provide calorie levels to the nearest 50 kcals (e.g., 1100 kcal, 1150 kcal, 1200 kcal, etc.). They are educated by the GCRC RDs and provided menus to guide their food purchasing and preparation of daily breakfast meals that are consistent with the prescribed calorie level. They are asked to consume only the food that is given to them or that is approved from the breakfast menu. All participants will pick up their food 3 times/wk during the intervention, and are asked to keep a log of everything they eat or drink.

Exercise intervention: The exercise will take place in an exercise facility at the Geriatric Research Center on the campus of the Wake Forest University/Baptist Medical Center. Two study personnel, including at least one trained technician, will supervise all exercise sessions. Emergency equipment will be kept on site during exercise sessions. Blood pressure and heart rate (HR) will be measured before each exercise session and subjects will warm-up by walking for 3-5 min at a slow pace and will then walk at an intensity of 65-70% of heart rate reserve (HRR, assessed during the VO2max test). The duration of walking exercise will progress from 15-20 mins at 50% HRR the 1st week to 30 mins at 65-70% HRR by the end of the 6th week and thereafter. Each walking session will end with a 3-5 min cool-down followed by 5 min of large muscle flexibility exercise.

ELIGIBILITY:
Inclusion Criteria:

* BMI=30-34.9 kg/m2
* Sedentary for past 6 months (<30 min, 3 d/wk of exercise, including walking)
* Normal cognitive function (MMSE >24)
* No contraindications for participation in weight loss or exercise (e.g., severe arthritis or musculoskeletal disorders)
* Able to provide own transportation to study visits and intervention
* No drug abuse or excessive alcohol use (> 7 drinks/week)
* Not dependent on a cane or walker

Exclusion Criteria:

* Weight loss or gain (±5%) in past 6 months
* Body weight >136.4 kg (DXA limit is 300 lbs)
* Smoker (No nicotine within past year)
* Osteoporosis (T-score ≥ -2.5)
* Abnormal kidney function tests
* Insulin-dependent or uncontrolled diabetes
* Uncontrolled hypertension (BP>200/110 mmHg)
* Hypertriglyceridemia (TG>400 mg/dl)
* Past or current ischemic heart disease, angina, heart failure, peripheral artery disease, stroke, chronic respiratory disease, uncontrolled endocrine/metabolic disease, neurological or hematological disease, clinically evident edema
* Cancer requiring treatment in past 2 years, except non-melanoma skin cancers
* Severe anemia (Hb<10 g/100 ml)
* Hip fracture, hip or knee replacement, or spinal surgery in past 6 months
* Regular use of medications that influence study variables (growth/steroid hormones, estrogen, anti-inflammatory, beta blockers, etc.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 180 (Actual)
Dates: Start 2009-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
maximal aerobic capacity (VO2max) and functional endurance (400 m walk time) | assessment visits will take place at baseline and post 5 months intervention

SECONDARY OUTCOMES:
changes in specific CVD risk factors (inflammatory markers, blood lipids, blood pressure, and glucose tolerance) | baseline and 5-month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Wake Forest University, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Brinkley TE, Leng I, Bailey MJ, Houston DK, Hugenschmidt CE, Nicklas BJ, Hundley WG. Effects of Exercise and Weight Loss on Proximal Aortic Stiffness in Older Adults With Obesity. Circulation. 2021 Aug 31;144(9):684-693. doi: 10.1161/CIRCULATIONAHA.120.051943. Epub 2021 Aug 2. PMID 34333991